CLINICAL TRIAL: NCT03878810
Title: Effects of Video Game-based Physical Activity Training in Persons With Multiple Sclerosis With Restless Legs Syndrome
Brief Title: Exergaming in Persons With Multiple Sclerosis With Restless Legs Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/01-138
Record Dates: First submitted 2019-02-04; First posted 2019-03-18 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exergaming, restless legs syndrome (+) (Experimental): A video game-based physical activity training will be applied under a physiotherapist supervision for 2 days/week for 8 weeks.
  Interventions: Behavioral: Exergaming
- Exergaming, restless legs syndrome (-) (Experimental): A video game-based physical activity training will be applied under a physiotherapist supervision for 2 days/week for 8 weeks.
  Interventions: Behavioral: Exergaming
- Control, restless legs syndrome (+) (No Intervention): No specific intervention.
- Control, restless legs syndrome (-) (No Intervention): No specific intervention.

INTERVENTIONS:
Behavioral: Exergaming — A video game-based physical activity training applied using a commercial game console.
  Arms: Exergaming, restless legs syndrome (+); Exergaming, restless legs syndrome (-)

SUMMARY:
In this studly, the effects of an 8-week videogame-based physical activity training in persons with multiple sclerosis will be investigated.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic, progressive, and demyelinating disease of the central nervous system that affects more than 2.5 million people worldwide and is more common in young adults. The most common clinical signs and symptoms include fatigue, spasticity, cognitive impairment, chronic pain, depression, decreased quality of life, and bladder and bowel dysfunction.

Sleep disturbance is affecting more than 50% of persons with multiple sclerosis. Restless legs syndrome is one of the factors causing sleep disturbance in persons with multiple sclerosis. Studies have showed that the incidence of restless legs syndrome in persons with multiple sclerosis is about five times more than the general population.

In order to increase and maintain the quality of life of persons with multiple sclerosis, the disease-related progressive symptoms need to be managed. Therefore, persons with multiple sclerosis need long-term rehabilitation. This situation reduces the motivation of the people over time and makes the continuity of treatment difficult. Developments in rehabilitation technology aim to contribute to the treatment process as well as to increase the active participation of individuals with chronic diseases.

Current literature has shown that video-based physical activity training as non-pharmacological therapy may be an effective method for symptoms such as balance, walking, fatigue, cognitive functions in persons with multiple sclerosis, but the effects on restless legs syndrome are not known.

The main aim of the study is to investigate the effects of 8-week video game-based physical activity training in persons with multiple sclerosis with restless legs syndrome.

Persons who followed by the outpatient Multiple Sclerosis Clinic of Dokuz Eylül University Hospital will participate in the study. A total of 68 participants will randomly be divided into 4 groups as exergaming group and control group with restless legs syndrome, exergaming group and control group without restless legs syndrome.

A video game-based physical activity training will apply to exergaming groups by a physiotherapist for 2 days/week. The control groups will continue their routine treatment during the study. After the study, the treatment options will be offered to the participants. Assessments will done at baseline, after 8 weeks (post-treatment) and at 8 weeks (follow-up). Assessments will be done by assessors who are blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* A relapsing-remitting or secondary progressive type of multiple sclerosis,
* Being able to walk at least 100 meters without resting,
* Being able to stably stand for half an hour,
* To be willing to participate in the study.

Exclusion Criteria:

* Another neurological disorder,
* Relapse during the study period,
* Orthopedic surgery history including the ankle-foot, knee, hip, or spine, affecting balance,
* Diagnosed severe cognitive and/or psychiatric impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group rating scale for restless legs syndrome | Change from Baseline at 8 and 16 weeks
  The International Restless Legs Syndrome Study Group rating scale for restless legs syndrome is used to assess severity of the restless legs syndrome symptoms. It consists of 10 items scored by 0 to 4. Possible scores range from 0 to 40. Higher scores indicate higher severity.

SECONDARY OUTCOMES:
Timed 25-Foot Walk | Change from Baseline at 8 and 16 weeks
  The Timed 25-Foot Walk is a quantitative mobility and leg function performance test based on a timed 25-walk. he patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score is the average of the two completed trials. Higher time represents slower walking speed and more walking impairment.
12-Item Multiple sclerosis walking scale | Change from Baseline at 8 and 16 weeks
  The 12-Item Multiple sclerosis walking scale is a self-assessment scale which measures the impact of multiple sclerosis on walking. It consists of 12 questions with Likert-type choose options concerning the limitations to walking due to multiple sclerosis during the past 2 weeks. Total score ranges 0 from 100. Higher scores indicate more impact of multiple sclerosis on walking.
Modified Fatigue Impact Scale | Change from Baseline at 8 and 16 weeks
  The Modified Fatigue Impact Scale provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The scale consists of 21 items with a Likert-type choose options. The total score for the scale is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items. The total score ranges from 0 to 84. Higher score indicates higher level of fatigue.
Timed Up and Go test | Change from Baseline at 8 and 16 weeks
  The Timed Up and Go test is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require. The time is calculated from the initiation of the instruction to start and ends when the patient has sit down. Higher time represents more static and dynamic balance and mobility impairment.
6-Minute Walk Test | Change from Baseline at 8 and 16 weeks
  The 6-Minute Walk Test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The goal is for the individual to walk as far and fast as possible in 6 minutes. The total distance is recorded. Higher distance represents a better submaximal exercise capacity.
Epworth Sleepiness Scale | Change from Baseline at 8 and 16 weeks
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Godin Leisure Time Exercise Questionnaire | Change from Baseline at 8 and 16 weeks
  The Godin Leisure Time Exercise Questionnaire is a commonly used questionnaire to measure of usual physical activity in persons with multiple sclerosis. It contains three items that measure the frequency of strenuous, moderate, and mild physical activities for periods of more than 15 minutes during one's free time within a typical week. Weekly frequencies of strenuous, moderate and mild physical activity were multiplied by 9, 5 and 3 metabolic equivalents, respectively, and were summed to form a measure of the total leisure physical activity. Higher scores indicate higher level of physical activity.
Hospital Anxiety And Depression Scale - Anxiety | Change from Baseline at 8 and 16 weeks
  The scale aims to measure symptoms of generalized anxiety disorder and consists of 7 items, seven items. Each item is scored on a response-scale with four alternatives ranging between 0 and 3. Higher scores indicate higher symptoms.
Hospital Anxiety And Depression Scale - Depression | Change from Baseline at 8 and 16 weeks
  The scale aims to measure symptoms of depression and consists of 7 items, seven items. Each item is scored on a response-scale with four alternatives ranging between 0 and 3. Higher scores indicate higher symptoms.
Multiple Sclerosis International Quality of Life questionnaire | Change from Baseline at 8 and 16 weeks
  The Multiple Sclerosis International Quality of Life questionnaire is a disease-specific, self-administered, multidimensional questionnaire, was co-developed and initially validated in 15 countries including Turkey. The questionnaire comprises 31 questions in 9 subscales: activities of daily living, psychological well-being, symptoms, relationships with friends, relationships with family, sentimental and sexual life, coping, rejection, and relationships with healthcare system. All 9 dimensions and the index score were linearly transformed and standardized on a 0-100 scale, where 0 indicates the worst possible level of quality of life and 100 indicates the best level.
Multiple Sclerosis-Related Symptom Checklist | Change from Baseline at 8 and 16 weeks
  Multiple Sclerosis-Related Symptom Checklist has 26 items that consist 5 subsections and 2 independent items. Sub-sections evaluate motor (7 items), brainstem (4 items), sensory (4 items), neuropsychiatric problems (3 items) and excretory problems (6 items). Independent items are related with fatigue and sleep difficulty. Responses are in the form of a 6-point Likert scale (None: 0, almost no: 1, sometimes: 2, usually: 3, almost always: 4, always: 5). The minimum score that can be taken from the scale is 0, the maximum score is 130, and the high score shows an increased symptom load.

OTHER OUTCOMES:
Restless Legs Syndrome Diagnostic Criteria | At Baseline
  Diagnostic Criteria for Restless Legs Syndrome was developed by the Restless Legs Syndrome Working Group in 1995 and revised in 2003 and 2014. These criteria include; the need to move the legs due to uncomfortable or unpleasant sensations in the legs, the need for movement or disturbing sensations start or worsen at rest, the need for movement or disturbing sensations can be partially or totally relieved by movements such as walking or stretching, the need for movement or disturbing sensations may worsen at night or only occur in the evening or night, The aforementioned features cannot be considered only in relation to primary symptoms or other medical or behavioral conditions (e.g., myalgia, venous stasis, leg edema, leg cramps, habitual foot swing). Patients meeting all of the criteria are diagnosed with restless legs syndrome. The restless legs syndrome diagnosis will be confirmed by a neurologist.
Expanded Disability Status Scale | At Baseline
  The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale is based on a neurological examination by a clinician. It has steps from 0 to 10. The higher scores indicate higher neurological disability.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Ozakbas, MD, Study Director — Izmir Katip Celebi University
Locations (1):
- MS Outpatient Clinic, Dokuz Eylul University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided